CLINICAL TRIAL: NCT06421714
Title: A Phase I, Single-Center, Open-Label, Two-Period, Single Sequence, Two Treatment Drug-Drug Interaction Study of GZ/SAR402671 (Venglustat) and Itraconazole in Healthy Male Subjects
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of Orally Administered Venglustat and Itraconazole in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT14339; 2014-002550-39 (EudraCT Number)
Record Dates: First submitted 2024-05-13; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — venglustat; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venglustat and Itraconazole (Experimental): The first period will include a single dose administration of venglustat followed by a second period including a multiple dose administration of itraconazole for 12 days and a second single dose administration of venglustat on the 6th day of itraconazole administration
  Interventions: Drug: Venglustat; Drug: Itraconazole

INTERVENTIONS:
Drug: Venglustat — Pharmaceutical form:Capsule-Route of administration:Oral
  Other Names: GZ/SAR402671
Drug: Itraconazole — Pharmaceutical form:Capsule-Route of administration:Oral
  Other Names: ITZ; Sporanox

SUMMARY:
The purpose of this study is to assess in healthy adult male participants the effects of itraconazole on the pharmacokinetics of venglustat and to assess the safety and tolerability of venglustat with and without coadministration of itraconazole. The maximum duration for participants from screening is between 32 to 62 days.

DETAILED DESCRIPTION:
Total study duration for participants is up to 62 days including screening up to 28 days, 1 day of treatment in period 1, washout of 7 days, 13 days of treatment in period 2, and follow up period 10-14 days after last dose.

ELIGIBILITY:
Inclusion Criteria: -Male participants, between 18 and 55 years of age, inclusive.

* Body weight between 50.0 and 100.0 kg, inclusive, body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs, electrocardiogram, and laboratory parameters.
* Having given written informed consent prior to undertaking any study-related procedure.
* Not under any administrative or legal supervision.
* Male participant, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom) plus (spermicide or intra-uterine device or hormonal contraceptive) from the inclusion up to 4 months after the last dosing.
* Male participant, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 4 months after the last dosing.
* Male participant has agreed not to donate sperm from the inclusion up to 4 months after the last dosing. Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension excluding vasovagal episode associated with a blood draw.
* Presence or history of clinically significant drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* Smoking regularly more than 5 cigarettes or equivalent per week, unable to stop smoking during the study (occasional smoker can be enrolled). Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency Virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen or urine alcohol test.
* Any contraindications to itraconazole, according to the applicable labeling.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of venglustat | Multiple time points up to 21 days
Area under the plasma concentration versus time curve calculated from time zero to the real time (tlast) (AUClast) of venglustat | Multiple time points up to 21 days

SECONDARY OUTCOMES:
Maximum plasma concentration observed (Cmax) of venglustat | Multiple time points up to 21 days
Plasma concentration observed just before treatment administration during repeated dosing (Ctrough) of venglustat | Multiple time points up to 21 days
Time to reach Cmax (tmax) of venglustat | Multiple time points up to 21 days
Terminal half-life (t1/2) of venglustat | Multiple time points up to 21 days
Maximum plasma concentration observed (Cmax) of itraconazole | Multiple time points up to 21 days
Plasma concentration observed just before treatment administration during repeated dosing (Ctrough) of itraconazole | Multiple time points up to 21 days
Time to reach Cmax (tmax) of itraconazole | Multiple time points up to 21 days
Area under the plasma concentration versus time curve calculated over the dosing interval (12 h) (AUC0-12) of itraconazole | Multiple time points up to 21 days
Maximum plasma concentration observed (Cmax) of hydroxyitraconazole | Multiple time points up to 21 days
Plasma concentration observed just before treatment administration during repeated dosing (Ctrough) of hydroxyitraconazole | Multiple time points up to 21 days
Time to reach Cmax (tmax) of hydroxyitraconazole | Multiple time points up to 21 days
Area under the plasma concentration versus time curve over the dosing interval (12 h) (AUC0-12) of hydroxyitraconazole | Multiple time points up to 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org